CLINICAL TRIAL: NCT00888082
Title: Protection of Ovarian Function With Goserelin Acetate in Premenopausal Early Breast Cancer Patients Undergoing Adjuvant Chemotherapy: An Open Label, Randomised, Multi-Centre, Phase IIIb Study
Brief Title: Protection of Ovarian Function With Goserelin Acetate in Premenopausal Early Breast Cancer Patients With Chemotherapy
Acronym: PROOF
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: MC MD, AstraZeneca Pharmaceuticals
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: D8664L00012
Record Dates: First submitted 2009-04-23; First posted 2009-04-24 (Estimated); Last update posted 2010-12-10 (Estimated); Status verified 2010-12

CONDITIONS: Breast Cancer; Ovarian Function
Keywords: adjuvant chemotherapy; breast cancer; goserelin acetate; ovarian function; Chemotherapy; Primary invasive breast cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Goserelin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- A (No Intervention): Patients receiving only adjuvant chemotherapy
- B (Experimental): Patient receiving goserelin acetate along with adjuvant chemotherapy
  Interventions: Drug: Goserelin acetate

INTERVENTIONS:
Drug: Goserelin acetate — 3.6 mg depot injectable preparation
  Other Names: Zoladex 3.6 mg Depot
  Arms: B

SUMMARY:
Primary objective of this study is to determine the effectiveness of goserelin acetate (Zoladex) in preserving ovarian function in premenopausal women undergoing adjuvant chemotherapy for primary invasive breast cancer by documenting persistence or resumption of regular menses via menstrual history, serum FSH and E2 measurements.

The secondary objectives of this study are as follows: To investigate the impact of treatment with chemotherapy with or without goserelin acetate (i.e. impact of the expectation of ovarian function preservation) on participants' quality of life (QOL) by FACT-ES scale, and to compare safety and tolerability of study drugs in two treatment groups by evaluation of adverse events.

ELIGIBILITY:
Inclusion Criteria:

* Pathologically confirmed invasive breast carcinoma
* Candidates for adjuvant chemotherapy for primary breast cancer
* Premenopausal, verified before chemotherapy is begun as satisfying both cyclic vaginal bleeding and appropriate hormone levels

Exclusion Criteria:

* Previous systemic chemotherapy
* Pregnancy
* Stage IV breast cancer

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 102 (Estimated)
Dates: Primary Completion 2012-04 (Estimated); Study Completion 2012-04 (Estimated)

PRIMARY OUTCOMES:
The ovarian function will be considered as regained, if E2 measurements return to premenopausal levels (equal to or above 20 pg/ml), FSH measurements return to premenopausal levels (less than or equal to 40 IU/L) | Each 3 months
The ovarian function will be considered as regained, if menstrual bleeding is observed in two consecutive menstrual cycles | Each 3 months

SECONDARY OUTCOMES:
Quality of life (QOL) through-out the study measured by FACT-ES scale. | Each 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Mustafa Özgüroğlu, Assoc.Prof., Study Chair — Istanbul University Cerrahpasa Medical Faculty, Medical Oncology Clinic, Cerrahpasa 34098, Istanbul, Turkey; Yeşim Eralp, Assoc.Prof., Principal Investigator — Istanbul University Istanbul Medical Faculty, Oncology Institute, Medical Oncology Department, Capa 34360 Istanbul, Turkey; Gül Başaran, Assoc.Prof., Principal Investigator — Marmara University Medical Faculty, Medical Oncology Department, Istanbul, Turkey; Kadri Altundağ, Prof., Principal Investigator — Hacettepe University Medical Faculty, Medical Oncology Department, Sihhiye 06100 Ankara, Turkey; Filiz Çay Şenler, Assoc.Prof., Principal Investigator — Ankara University Medical Faculty, Medical Oncology Department, Sihhiye 06100 Ankara, Turkey; Metin Özkan, Principal Investigator — Erciyes University Medical Faculty, Medical Oncology Department, 38039 Kayseri, Turkey
Locations (3):
- Turkey (Türkiye) (3):
  - Research Site, Ankara
  - Research Site, Istanbul
  - Research Site, Kayseri

REFERENCES:
- [Background] Ataya K, Rao LV, Lawrence E, Kimmel R. Luteinizing hormone-releasing hormone agonist inhibits cyclophosphamide-induced ovarian follicular depletion in rhesus monkeys. Biol Reprod. 1995 Feb;52(2):365-72. doi: 10.1095/biolreprod52.2.365. PMID 7711205
- [Background] Ataya KM, McKanna JA, Weintraub AM, Clark MR, LeMaire WJ. A luteinizing hormone-releasing hormone agonist for the prevention of chemotherapy-induced ovarian follicular loss in rats. Cancer Res. 1985 Aug;45(8):3651-6. PMID 3926307
- [Background] Bines J, Oleske DM, Cobleigh MA. Ovarian function in premenopausal women treated with adjuvant chemotherapy for breast cancer. J Clin Oncol. 1996 May;14(5):1718-29. doi: 10.1200/JCO.1996.14.5.1718. PMID 8622093
- [Background] Blumenfeld Z, Eckman A. Preservation of fertility and ovarian function and minimization of chemotherapy-induced gonadotoxicity in young women by GnRH-a. J Natl Cancer Inst Monogr. 2005;(34):40-3. doi: 10.1093/jncimonographs/lgi015. PMID 15784821
- [Background] Bokser L, Szende B, Schally AV. Protective effects of D-Trp6-luteinising hormone-releasing hormone microcapsules against cyclophosphamide-induced gonadotoxicity in female rats. Br J Cancer. 1990 Jun;61(6):861-5. doi: 10.1038/bjc.1990.192. PMID 2142603
- [Background] Brincker H, Rose C, Rank F, Mouridsen HT, Jakobsen A, Dombernowsky P, Panduro J, Andersen KW. Evidence of a castration-mediated effect of adjuvant cytotoxic chemotherapy in premenopausal breast cancer. J Clin Oncol. 1987 Nov;5(11):1771-8. doi: 10.1200/JCO.1987.5.11.1771. PMID 3316514
- [Background] Cheer SM, Plosker GL, Simpson D, Wagstaff AJ. Goserelin: a review of its use in the treatment of early breast cancer in premenopausal and perimenopausal women. Drugs. 2005;65(18):2639-55. doi: 10.2165/00003495-200565180-00011. PMID 16392882
- [Background] Del Mastro L, Catzeddu T, Boni L, Bell C, Sertoli MR, Bighin C, Clavarezza M, Testa D, Venturini M. Prevention of chemotherapy-induced menopause by temporary ovarian suppression with goserelin in young, early breast cancer patients. Ann Oncol. 2006 Jan;17(1):74-8. doi: 10.1093/annonc/mdj029. Epub 2005 Oct 27. PMID 16254024
- [Background] Del Mastro L, Venturini M, Sertoli MR et al. Phase III adjuvan trial comparing standard versus accelerated FEC regimen in early breast cancer patients. Results from GONO-MIG1 study. Breast Cancer Res Treat 2003; 82 (Suppl 1): S9 (Abstr).
- [Background] Del Mastro L, Venturini M, Sertoli MR, Rosso R. Amenorrhea induced by adjuvant chemotherapy in early breast cancer patients: prognostic role and clinical implications. Breast Cancer Res Treat. 1997 Apr;43(2):183-90. doi: 10.1023/a:1005792830054. PMID 9131274
- [Background] Polychemotherapy for early breast cancer: an overview of the randomised trials. Early Breast Cancer Trialists' Collaborative Group. Lancet. 1998 Sep 19;352(9132):930-42. PMID 9752815